CLINICAL TRIAL: NCT05569252
Title: A Phase 2, 12-Week, Randomized, Double-Blind, Placebo-Controlled Study of DS-1211b in Individuals With PseudoXanthoma Elasticum
Brief Title: A Study of DS-1211b in Individuals With PseudoXanthoma Elasticum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: PXE International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS1211-A-U201; 2022-000676-19 (EudraCT Number)
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Pseudoxanthoma Elasticum
Keywords: Pseudoxanthoma Elasticum; DS-1211b
MeSH Terms: conditions — Pseudoxanthoma Elasticum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DS-1211b low dose (Experimental): Participants who will be randomized to receive a DS-1211 tablet once daily for 12 weeks.
  Interventions: Drug: DS-1211b
- DS-1211b middle dose (Experimental): Participants who will be randomized to receive a DS-1211b tablet once daily for 12 weeks.
  Interventions: Drug: DS-1211b
- DS-1211b high dose (Experimental): Participants who will be randomized to receive a DS-1211b tablet once daily for 12 weeks.
  Interventions: Drug: DS-1211b
- Placebo (Placebo Comparator): Participants who will be randomized to receive a placebo tablet once daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DS-1211b — DS-1211b tablet administered once daily in the morning either in the fasted state or with a meal
  Arms: DS-1211b high dose; DS-1211b low dose; DS-1211b middle dose
Other: Placebo — Placebo tablet administered once daily in the morning either in the fasted state or with a meal
  Arms: Placebo

SUMMARY:
This study was designed to evaluate the safety, tolerability, pharmacodynamics (PD) of DS-1211b, and pharmacokinetics (PK) in individuals with Pseudoxanthoma elasticum (PXE). PXE is a rare disease that is associated with significant risks of visual impairments and comorbidity from peripheral and cardiovascular diseases, and adversely impacts the quality of life in afflicted individuals.

DETAILED DESCRIPTION:
DS-1211b, a potent small-molecule inhibitor of tissue-nonspecific alkaline phosphatase, is being developed for the treatment ectopic calcification diseases such as PXE. This study will assess DS-1211b (low-, middle-, and high-dose tablets) administered once daily for 12 weeks in individuals with PXE.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed and dated informed consent
* Male or female participants aged 18 to 75 years at screening
* Have an established diagnosis of PXE
* Fully vaccinated for coronavirus disease 2019 (COVID-19) per current Center for Disease Control and Prevention guidelines

Key Exclusion Criteria:

* Have a history of bone fracture in the past 6 months
* Have a history of active metabolic bone disease, excluding osteopenia or osteoporosis without fragility fracture
* Have a history of calcium pyrophosphate deposit disease
* Have a history of hypophosphatasia
* Have a history of untreated hyperparathyroidism
* Participated in another interventional research study in the past 60 days.
* Used bisphosphonate in the preceding 12 months or had plans to use bisphosphonate during the study.
* Received Vitamin B6 supplementation >5 mg/day in the month prior to screening and during the study
* Initiated or changed dose of Vitamin D in the preceding month prior to screening
* Have an alkaline phosphatase <lower limit of normal (LLN) range
* Have a QTcF interval duration >450 ms at screening
* Have moderate to severe renal insufficiency
* Are pregnant or breast-feeding women
* Are female participants unwilling to use contraceptive methods
* Have any elective surgery planned during the study period
* Have any other significant condition (medical, psychiatric, social, or medication) that, in the judgment of the Investigator, would prevent full participation or would be inappropriate for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Daiichi Sankyo
Locations (7):
- United States (6):
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Boston Neuro Research Center, North Dartmouth, Massachusetts
  - Infinity Medical Research Inc, North Dartmouth, Massachusetts
  - Frontage Clinical Services, Inc., Secaucus, New Jersey
  - Clinilabs, New York, New York
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 65 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study in the United States and in the Netherlands.
Groups:
- DS-1211b Low Dose: Participants who were randomized to receive DS-1211 tablets once daily for 12 weeks.
- DS-1211b Middle Dose; DS-1211b High Dose: Participants who were randomized to receive DS-1211b tablets once daily for 12 weeks.
- Placebo: Participants who were randomized to receive placebo tablets once daily for 12 weeks.
Period: Overall Study
Arm/Group | DS-1211b Low Dose | DS-1211b Middle Dose | DS-1211b High Dose | Placebo
Started | 16 | 16 | 16 | 17
Completed | 15 | 16 | 16 | 17
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse event (central vision loss) | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographics and baseline characteristics were assessed in the Intent-to-Treat Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | DS-1211b Low Dose | DS-1211b Middle Dose | DS-1211b High Dose | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 16 | 17 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (7.65) | 51.6 (10.84) | 53.8 (8.47) | 53.5 (13.92) | 53.7 (10.43)
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 14 | 12 | 54
  ≥64 years | 2 | 2 | 2 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 10 | 14 | 41
  Male | 9 | 6 | 6 | 3 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 16 | 15 | 16 | 16 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) in Participants Receiving DS-1211b
Description: TEAEs are defined as events that start on or after the first dose of study drug or start prior to but then worsen after the first dose of study drug. Adverse events are coded using MedDRA version 26.1.
Time Frame: From the date of signing informed consent form up to Day 98 (14 days after last dose of study drug) post-dose of 12-week treatment period
Population: Treatment-emergent adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1211b Low Dose | DS-1211b Middle Dose | DS-1211b High Dose | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 17
Participants
  Any TEAE | 8 | 7 | 6 | 6
  Any TEAE leading to death | 0 | 0 | 0 | 0
  Any TEAE by maximum severity, mild | 4 | 6 | 4 | 3
  Any TEAE by maximum severity, moderate | 3 | 1 | 2 | 3
  Any TEAE by maximum severity, severe | 1 | 0 | 0 | 0
  Any serious TEAE | 1 | 0 | 0 | 0
  Any serious TEAE leading to drug interruption | 0 | 0 | 0 | 0
  Any serious TEAE leading to drug discontinuation | 0 | 0 | 0 | 0
  Any serious TEAE related to study drug | 0 | 0 | 0 | 0
  Any TEAE leading to drug interruption | 1 | 0 | 0 | 0
  Any TEAE leading to drug discontinuation | 1 | 0 | 0 | 0
  Any TEAE related to study drug | 2 | 2 | 1 | 1
  Any related TEAE leading to drug interruption | 1 | 0 | 0 | 0
  Any related TEAE leading to drug discontinuation | 1 | 0 | 0 | 0
  Any TEAE related to COVID-19 | 0 | 0 | 1 | 1

2. Primary Outcome: Percent Change From Baseline in Pharmacodynamic Parameter Alkaline Phosphatase (ALP) Levels
Description: ALP levels were assessed using the IFCC serum assay.
Time Frame: Pre-dose on Days 15, 43, 84; Day 86-88 and Day 98 of 12-week treatment period
Population: ALP levels were assessed in participants with available data in the Biomarker Analysis Set.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DS-1211b Low Dose | DS-1211b Middle Dose | DS-1211b High Dose | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 17
percent change
  Day 15: number analyzed (Participants) | 16 | 16 | 16 | 15
  Day 15 | 17.93 (10.60) | 24.39 (14.45) | 39.40 (11.52) | -0.48 (6.14)
  Day 43: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 43 | 25.02 (17.54) | 42.89 (30.26) | 63.48 (35.68) | -2.54 (10.38)
  Day 84: number analyzed (Participants) | 15 | 16 | 16 | 16
  Day 84 | 25.54 (16.89) | 39.81 (20.19) | 61.90 (37.86) | -4.31 (9.58)
  Day 86-88: number analyzed (Participants) | 15 | 15 | 13 | 16
  Day 86-88 | 16.60 (18.39) | 29.93 (14.61) | 49.67 (26.00) | -3.20 (9.46)
  Day 98: number analyzed (Participants) | 14 | 15 | 13 | 17
  Day 98 | 7.65 (15.34) | 9.48 (14.99) | 22.95 (22.42) | -0.05 (13.72)

3. Primary Outcome: Percent Change From Baseline in Pharmacodynamic Parameter Inorganic Pyrophosphate (PPi) Levels
Description: PPi levels were assessed from collected plasma.
Time Frame: Pre-dose on Days 15, 43, and 84 of 12-week treatment period
Population: PPi levels were assessed in participants with available data in the Biomarker Analysis Set.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DS-1211b Low Dose | DS-1211b Middle Dose | DS-1211b High Dose | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 17
percent change
  Day 15 | 118.97 (362.42) | 11.32 (50.13) | 23.95 (69.94) | 13.33 (61.00)
  Day 43: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 43 | 17.75 (50.05) | -5.55 (36.74) | 4.59 (19.47) | 12.97 (38.33)
  Day 84: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 84 | 23.48 (78.04) | 81.77 (313.08) | 24.27 (97.87) | 4.28 (41.45)

4. Primary Outcome: Percent Change From Baseline in Pharmacodynamic Parameter Pyridoxal 5'-Phosphate (PLP) Levels
Description: PLP levels were assessed from collected plasma.
Time Frame: Pre-dose on Days 15, 43, 84; Day 86-88 and Day 98 of 12-week treatment period
Population: PLP levels were assessed using Biomarker Analysis Set.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DS-1211b Low Dose | DS-1211b Middle Dose | DS-1211b High Dose | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 17
percent change
  Day 15 | 11.01 (53.93) | 45.42 (92.18) | 50.97 (56.78) | 3.42 (36.86)
  Day 43: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 43 | 8.56 (42.26) | 36.73 (79.89) | 25.00 (48.51) | 16.25 (35.09)
  Day 84: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 84 | 12.03 (46.95) | 53.07 (110.74) | 6.04 (38.72) | -8.44 (41.44)
  Day 86-88: number analyzed (Participants) | 14 | 14 | 13 | 16
  Day 86-88 | -5.96 (27.93) | -6.52 (41.25) | -28.76 (31.72) | -10.77 (45.53)
  Day 98: number analyzed (Participants) | 14 | 14 | 16 | 17
  Day 98 | 6.10 (47.54) | -10.96 (45.58) | -8.41 (35.10) | 17.07 (98.34)

5. Secondary Outcome: Pharmacokinetic Parameter Maximum Concentration (Cmax)
Description: Pharmacokinetic parameter Cmax was estimated using population PK modeling.
Time Frame: Day1 and Day 84 post-dose of 12-week treatment period
Population: Pharmacokinetic parameters were assessed using PK Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DS-1211b Low Dose | DS-1211b Middle Dose | DS-1211b High Dose
Number analyzed (Participants) | 16 | 16 | 16
ng/mL
  Day 1 | 252 (20.5) | 540 (34.8) | 713 (26.9)
  Day 84 | 255 (20.6) | 547 (34.9) | 726 (27.0)

6. Secondary Outcome: Pharmacokinetic Parameter Time to Maximum Concentration (Tmax)
Description: Pharmacokinetic parameter Tmax was assessed using population PK modeling.
Time Frame: Day 1 and Day 84 post-dose of 12-week treatment period
Population: Pharmacokinetic parameters were assessed using PK Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | DS-1211b Low Dose | DS-1211b Middle Dose | DS-1211b High Dose
Number analyzed (Participants) | 16 | 16 | 16
hours
  Day 1 | 1.25 [0.75 to 2.00] | 1.13 [0.75 to 3.75] | 1.25 [0.75 to 1.75]
  Day 84 | 1.25 [0.75 to 2.00] | 1.13 [0.75 to 3.75] | 1.25 [0.75 to 1.75]

7. Secondary Outcome: Pharmacokinetic Parameter Trough Plasma Concentration (Ctrough)
Description: Pharmacokinetic parameter Ctrough was assessed using observed concentrations at 10 hours post-dose.
Time Frame: Day 1 and Day 84 post-dose of 12-week treatment period
Population: Pharmacokinetic parameters were assessed in participants with available data in the PK Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DS-1211b Low Dose | DS-1211b Middle Dose | DS-1211b High Dose
Number analyzed (Participants) | 16 | 16 | 16
ng/mL
  Day 1 (10 hour): number analyzed (Participants) | 15 | 16 | 16
  Day 1 (10 hour) | 17.15 (11.58) | 26.30 (13.71) | 48.43 (46.50)
  Day 84 (10 hour): number analyzed (Participants) | 15 | 16 | 16
  Day 84 (10 hour) | 15.19 (9.00) | 38.53 (30.45) | 54.48 (40.79)

8. Secondary Outcome: Pharmacokinetic Parameter Area Under the Plasma Concentration-time Curve (AUC)
Description: Pharmacokinetic parameter AUCtau was assessed using population PK modeling.
Time Frame: Day 1 and Day 84 post-dose of 12-week treatment period
Population: Pharmacokinetic parameters were assessed using the PK Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | DS-1211b Low Dose | DS-1211b Middle Dose | DS-1211b High Dose
Number analyzed (Participants) | 16 | 16 | 16
ng*h/mL
  Day 1, AUCtau | 978 (28.3) | 2090 (28.0) | 2780 (32.1)
  Day 84, AUCtau | 1020 (29.3) | 2210 (29.0) | 3000 (33.7)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the time of signing the informed consent form up to 14 (±5) days after the last dose of study medication, up to 98 days.
Arm/Group | DS-1211b Low Dose | DS-1211b Middle Dose | DS-1211b High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/16 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 8/16 | 7/16 | 6/16 | 6/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-1211b Low Dose (N=16) | DS-1211b Middle Dose (N=16) | DS-1211b High Dose (N=16) | Placebo (N=17)
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DS-1211b Low Dose (N=16) | DS-1211b Middle Dose (N=16) | DS-1211b High Dose (N=16) | Placebo (N=17)
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fascitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Ophthalmic migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Central vision loss (Eye disorders) | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 1 | 0
SARS CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT05569252/Prot_SAP_000.pdf